CLINICAL TRIAL: NCT03983785
Title: The Effect of Pilates and Elastic Taping on Balance and Postural Control in Early Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Evrim Goz, Principal investigator, Dokuz Eylul University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: DokuzEU
Record Dates: First submitted 2019-06-09; First posted 2019-06-12 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
Keywords: Pilates; Elastic Taping; Balance; Postural control; Early Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates (Experimental)
  Interventions: Other: Pilates
- Elastic Taping (Experimental)
  Interventions: Other: Elastic taping
- Wait List Control (No Intervention)

INTERVENTIONS:
Other: Pilates — In pilates group: Pilates training twice a week for 6 weeks.
  Other Names: Elastic Taping
  Arms: Pilates
Other: Elastic taping — Elastic taping group: Elastic taping application after the pilates training twice a week for 6 weeks Wait List
  Arms: Elastic Taping

SUMMARY:
The aim of this study was to compare the effects of pilates training and elastic taping on balance and postural control in early Parkinson's patients.

DETAILED DESCRIPTION:
The subjects were randomly divided into 3 groups as pilates, elastic taping and waiting list control group. Individuals were given 60-minute pilates training twice a week for 6 weeks. In addition to Pilates training, elastic taping was applied twice a week for postural correction of the back. Individuals were evaluated for balance and postural control before and after training. Evaluation of clinical balance with Berg Balance Scale and Trunk Impairment Scale; Stability Limits, Sits Up, Normal and Tandem Walking Tests were performed with NeuroCom Balance Master balance and performance system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Parkinson Disease
* Mini Mental Test Score≥24
* Modified Hoehn and Yahr Score≤2
* Ability to stand 1 minute independently
* Ability to walk 10 meters

Exclusion Criteria:

* Other orthopaedic, neurologic or visual disease which could affect ability of balance and walking
* Unstabl cardiovasvularly disease
* History of Surgery about Parkinson disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Balance | 7.5 months
  Walk Across Test were performed with Neurocom Balance Master System.
Postural control | 7.5 months
  Stability Limits Test was performed with Neurocom Balance Master System.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Goz, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed?term=%22Gait+%26+posture%22%5BJour%5D+AND+Falaki%5Bauthor%5D&cmd=detailssearch